CLINICAL TRIAL: NCT06969820
Title: Establishment and Evaluation of Standardized Clinical, Biological and Imaging Parameters to Assess the Response of LDRT in Heel Spur With Plantar Fasciitis
Acronym: HEALSPUR
Status: Not yet recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 25-65-B
Record Dates: First submitted 2025-04-07; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Calcaneal Spur
MeSH Terms: conditions — Heel Spur | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment Group: Radiotherapy with a guideline-compliant (Radiotherapy of benign diseases; specialist group-specific evidence-based S2e guideline of the German Society for Radio-Oncology (DEGRO)) single dose of 0.5 Gy (3.0 Gy total dose) over 3 weeks and, if pain persists, a second series with the same dosage at 12-week intervals.
  Interventions: Procedure: Low-dose Radiation Therapy (LDRT) using MRI-based imaging techniques

INTERVENTIONS:
Procedure: Low-dose Radiation Therapy (LDRT) using MRI-based imaging techniques — LDRT using MRI-based imaging techniques by developing an MRI imaging protocol, deep learning-based image enhancement and resolution increase.

SUMMARY:
The clinical picture of calcaneal spur with plantar fasciitis is a debilitating disease that is difficult to treat with conservative and interventional measures. Radiotherapy has shown very good therapeutic results in retrospective data, which need to be clinically confirmed both subjectively and in terms of image morphology in a prospective approach.

Primary objective of the study:

To demonstrate a clinical benefit of LDRT: improvement of pain, functionality and quality of life after LDRT

ELIGIBILITY:
Inclusion Criteria:

* Age > 39 years
* Typical clinical picture of plantar fasciitis for at least 3 months without associated trauma, other musculoskeletal co-morbidities or degenerative joint disease
* Patients with first-time application of LDRT to the affected joint
* Willingness to cooperate and accessibility of patients, especially geographical proximity, for treatment and follow-up
* Patients for whom LDRT is indicated independently of the study
* Karnofsky Index >70%

Exclusion Criteria:

* Achillodynia ("dorsal" calcaneal spur)
* Previous trauma to the foot (fracture, tendon rupture)
* Musculoskeletal comorbidities of the foot
* Acute infections/open wounds in the area of the tendon to be examined or other relevant damage to the tendon to be examined
* Local steroid injections into the tendon prior to the study
* Rheumatic or vascular diseases, lymphedema
* Patients with tumors
* Individuals of childbearing potential who do not use adequate contraceptive measures consistently during therapy
* Persistent drug, medication or alcohol abuse
* Patients who have already undergone radiotherapy for the treatment of cancer
* Patients with an increased risk of an MRI examination, including the presence of metal implants, pacemakers or claustrophobia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heel spurs experience pain and inflammation, as do those with plantar fasciitis, which often goes hand in hand with it.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Proof of clinical benefit of LDRT using pain scale | 36 months
  Visual analog scale: pain scale from 0-10 (0..no pain - 10..worst pain)
Proof of clinical benefit of LDRT using QoL | 36 months
  QoL: SF-8 (Short Form-8 Health Survey), scale from 0-100 (0..worst score - 100..best score)
Proof of clinical benefit of LDRT using Calcaneodynia score | 36 months
  Calcaneodynia score, scale from 0-100 (0..worst performance - 100..best performance)
Proof of clinical benefit of LDRT using AOFAS Hindfoot Scale | 36 months
  AOFAS Hindfoot Scale, Score ranges from 0 to 100, with healthy ankles receiving 100 points.
Proof of clinical benefit of LDRT using Roles and Maudsley Scale | 36 months
  Roles and Maudsley scale is a 4-point subjective assessment used to evaluate patient pain and limitations in daily activities following treatment. It ranges from 1 (excellent result, no symptoms) to 4 (poor result, symptoms identical or worse than before treatment).

SECONDARY OUTCOMES:
Proof of an objectifiable clinical benefit of LDRT using MRI-based imaging techniques by developing an MRI imaging protocol | 36 months
Correlation of subjective pain parameters with laboratory chemical examinations. | 36 months
Correlation of subjective pain parameters, gait analyses and tendon elasticity with inflammatory components in the patient serum. | 36 months
Correlation of immune cell subpopulations with disease severity by correlating them with MRI and laboratory findings. | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Translational Radiobiology, Universitätsklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No